CLINICAL TRIAL: NCT03377738
Title: Randomized Clinical Trial About the Effectiveness of the Spirometry Test as a Motivational Tool for Quitting Tobacco in Primary Care
Brief Title: Effectiveness of the Spirometry Test as a Motivational Tool for Quitting Tobacco in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: MurciaSalud (Other Government); Public Health Service, Murcia (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRISA II.EPOC-Tabaco
Record Dates: First submitted 2011-06-22; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Tobacco Cessation
Keywords: Spirometry; Primary care; Smoking Cessations
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- anti-smoking therapy (No Intervention): All patients will be given only an intervention for tobacco cessation which will depend on the individual's cessation phase
- anti-smoking therapy + spirometry (Experimental): All patients will be given an intervention for tobacco cessation which will depend on the individual's cessation phase. In addition, in this group will be given a spirometry test as a motivational element for dishabituation.
  Interventions: Diagnostic Test: spirometry

INTERVENTIONS:
Diagnostic Test: spirometry — All patients will be given an intervention for tobacco cessation which will depend on the individual's cessation phase and will be given a spirometry test as a motivational element for dishabituation.
  Arms: anti-smoking therapy + spirometry

SUMMARY:
The purpose of this study is analyze if spirometry is a motivational element for changes in the cessation phases of the tobacco habit, compared with not done spirometry.

DETAILED DESCRIPTION:
According to data from the last INE health survey carried out in 2006, 31.4% of males and 22.3 % of females smoked, in other words more than 26% of the population were smokers. In the Region of Murcia, according to the same Health Survey, the data are even higher than those of Spain, with figures for male smokers at 36.25% and 23.31% for women, with an overall prevalence rate of nearly 30%.

In light of these data, it is necessary to carry out intervention to help tobacco cessation and in this regard,the 98% of smokers trying to quit on their own without any specific support do not achieve their goal.

Interventions at Primary Care Consultations we have two useful tools at our disposal: One of these is brief advice It should be firm, understandable, individualized, verbal and direct. It should last between 3 and 5 minutes and be eminently positive, highlighting the advantages of becoming an ex-smoker. This intervention vs non intervention have an OR=1.69 (IC 95%1.45-1.98). The other intervention we have in an intensive. This includes providing systematic anti-tobacco advice accompanied by written documentation and psychological support as well as the follow-up of patients in their dishabituation process, with a periodicity which varies according to different studies, although to do this more time will have to be dedicated in the consultation.

As more intense intervention on these patients as efficacy obtained is higher, increasing abstinence rates significantly.

Appropriate interventions based on stage of change are based on the transtheoretical model of Prochaska and DiClemente. Smokers are at one stage or another in terms of lesser or greater degree of motivation to quit being closely related to the phases of abandonment of tobacco.

In addition to these tools, two other interventions have been studied which could be useful for increasing cessation rates. In this regard, a Cochrane review determined the efficiency of the evaluation of biomedical risks and different levels of assessment used as a cessation tool for quitting the tobacco habit. The information from eleven trials was analyzed and in three of them spirometry and co-oximetry were used as motivational elements for tobacco cessation. However, the results were inconclusive due to the heterogeneity of the studies, but concludes that it is possible to further improve the methodological quality of studies aimed at evaluating the effectiveness of biomedical risk assessment, including spirometry, as an aid to quit smoking. Other studies also seen as a considerable number of smokers get smoking quit after learning their spirometric results.

For all of these reasons, it is necessary to carry out interventions which help to encourage tobacco habit cessation and in this regard this study has been designed, in which it is intended to assess spirometry , as a motivational element in the phase of tobacco cessation.

ELIGIBILITY:
Inclusion Criteria:

* An active smoker
* Aged between 40 and 75 years
* No diagnosis of acute or chronic respiratory disease

Exclusion Criteria:

* Serious or terminal diseases
* Limiting osteoarticular diseases
* Serious mental diseases: Psychosis
* Serious depressive disorder
* Neurosis
* Addiction to drugs/alcohol
* Displaced patients (not habitual residents)
* Pregnancy
* Spirometry carried out for any reason in the year prior to inclusion in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
- Number of cessations of the tobacco habit (%) | 2-3 weeks, 3 month and 6 months
- Cessation phase of the tobacco habit (%) | 2-3 weeks, 3 month and 6 months

SECONDARY OUTCOMES:
Score on the Richmond test for assessing motivation to quit smoking. | 2-3 weeks, 3 month and 6 months
Fagerström test score to assess dependency. | 2-3 weeks, 3 month and 6 months
Carbon monoxide levels (CO) (co-oximetry). | 2-3 weeks, 3 month and 6 months
Anthropometric variables: weight, size and body mass index Exposure to tobacco: nº packets/day. | 2-3 weeks, 3 month and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: A Lopez-santiago, MD, Principal Investigator — Consejeria de sanidad y consumo, Direccion general de planificacion, ordenacion sanitaria y farmaceutica e investigacion.
Locations (1):
- Fundación para la Formación e Investigación Sanitarias de la Región de Murcia, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Instituto Nacional de Estadística INE. Encuesta Nacional de Salud 2006.
- [Background] Ruiz CA, Pinedo AR, Miranda JA, Bermudez JA. [Spanish Society of Pulmonology and Thoracic Surgery (SEPAR) annual campaign for 2007: the year for smoking prevention and control]. Arch Bronconeumol. 2007 Aug;43(8):423-4. doi: 10.1016/s1579-2129(07)60097-4. No abstract available. Spanish. PMID 17692241
- [Background] Saiz Martinez-Acitores I, Rubio Colavida J, Espiga Lopez I, Alonso de la Iglesia B, Blanco Aguilar J, Cortes Mancha M, Cabrera Ortega JD, Pont Martinez P, Saavedra Rodriguez JM, Toledo Pallares J. [National Action Plan for Prevention and Tobacco Control]. Rev Esp Salud Publica. 2003 Jul-Aug;77(4):441-73. No abstract available. Spanish. PMID 12945131
- [Background] Banegas JR, Diez Ganan L, Gonzalez Enriquez J, Villar Alvarez F, Rodriguez-Artalejo F. [Recent decrease in smoking-attributable mortality in Spain]. Med Clin (Barc). 2005 May 28;124(20):769-71. doi: 10.1157/13075847. Spanish. PMID 15927102
- [Background] Villalbi JR, Castillo A, Cleries M, Salto E, Sanchez E, Martinez R, Tresserras R, Vela E; Barcelona Group. Acute myocardial infarction hospitalization statistics: apparent decline accompanying an increase in smoke-free areas. Rev Esp Cardiol. 2009 Jul;62(7):812-5. doi: 10.1016/s1885-5857(09)72362-x. English, Spanish. PMID 19709517
- [Background] Fernandez E, Fu M, Pascual JA, Lopez MJ, Perez-Rios M, Schiaffino A, Martinez-Sanchez JM, Ariza C, Salto E, Nebot M; Spanish Smoking Law Evaluation Group. Impact of the Spanish smoking law on exposure to second-hand smoke and respiratory health in hospitality workers: a cohort study. PLoS One. 2009;4(1):e4244. doi: 10.1371/journal.pone.0004244. Epub 2009 Jan 23. PMID 19165321
- [Background] Martinez-Sanchez JM, Fernandez E, Fu M, Perez-Rios M, Lopez MJ, Ariza C, Pascual JA, Schiaffino A, Perez-Ortuno R, Salto E, Nebot M. Impact of the Spanish smoking law in smoker hospitality workers. Nicotine Tob Res. 2009 Sep;11(9):1099-106. doi: 10.1093/ntr/ntp107. Epub 2009 Jul 29. PMID 19640834
- [Background] Silagy C. Physician advice for smoking cessation. Cochrane Database Syst Rev. 2000;(2):CD000165. doi: 10.1002/14651858.CD000165. PMID 10796499
- [Background] Clinical Practice Guideline Treating Tobacco Use and Dependence 2008 Update Panel, Liaisons, and Staff. A clinical practice guideline for treating tobacco use and dependence: 2008 update. A U.S. Public Health Service report. Am J Prev Med. 2008 Aug;35(2):158-76. doi: 10.1016/j.amepre.2008.04.009. PMID 18617085
- [Background] Sanz Pozo B, de Miguel Diez J, Camarelles Guillem F. [Non-pharmacological methods in tobacco dishabituation]. Rev Clin Esp. 2004 Jan;204(1):37-9. doi: 10.1157/13056793. No abstract available. Spanish. PMID 14746762
- [Background] Kottke TE, Battista RN, DeFriese GH, Brekke ML. Attributes of successful smoking cessation interventions in medical practice. A meta-analysis of 39 controlled trials. JAMA. 1988 May 20;259(19):2883-9. doi: 10.1001/jama.259.19.2883. PMID 3367456
- [Background] Camarelles Guillem F, Salvador Llivina T, Ramon Torell JM, Cordoba Garcia R, Jimenez Ruiz C, Lopez Garcia-Aranda V, Villalbi Hereter JR, Planchuelo Santos MA, Sanchez Monfort J, Lopez de Santiago A. [Consensus on health assistance for smoking control in Spain]. Rev Esp Salud Publica. 2009 Mar-Apr;83(2):175-200. doi: 10.1590/s1135-57272009000200004. Spanish. PMID 19626247
- [Background] F. Marqués Molías, et al. Recomendaciones sobre el estilo de vida. Grupo de Educación para la Salud del PAPPS. actualizacion 2009. acceso (23/03/2011): http://www.papps.org/upload/file/08%20PAPPS%20ACTUALIZACION%202009.pdf
- [Background] Javier Mataix Sancho et al. Guia para el tratamiento del tabaquismo activo y pasivo. segunda edicion 2009. accesso (24/03/2011): http://www.papps.org/upload/file/publicaciones/Guia%20Tabaquismo2009.pdf.
- [Background] Martin Cantera C, Cordoba Garcia R, Jane Julio C, Nebot Adell M, Galan Herrera S, Aliaga M, Pujol Ribera E, Ballestin M. [Mid-term evaluation of a help program for smokers]. Med Clin (Barc). 1997 Nov 29;109(19):744-8. Spanish. PMID 9470183
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Prochaska JO, Velicer WF, DiClemente CC, Fava J. Measuring processes of change: applications to the cessation of smoking. J Consult Clin Psychol. 1988 Aug;56(4):520-8. doi: 10.1037//0022-006x.56.4.520. No abstract available. PMID 3198809
- [Background] Bize R, Burnand B, Mueller Y, Rege Walther M, Cornuz J. Biomedical risk assessment as an aid for smoking cessation. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD004705. doi: 10.1002/14651858.CD004705.pub3. PMID 19370604
- [Background] Clotet J, Gomez-Arbones X, Ciria C, Albalad JM. [Spirometry is a good method for detecting and monitoring chronic obstructive pulmonary disease in high-risk smokers in primary health care]. Arch Bronconeumol. 2004 Apr;40(4):155-9. doi: 10.1016/s1579-2129(06)60207-3. Spanish. PMID 15030729
- [Background] Czajkowska-Malinowska M, Nowinski A, Gorecka D, Zielinski J. [Effects of spirometric screening in the community on smoking cessation]. Pneumonol Alergol Pol. 2001;69(9-10):524-9. Polish. PMID 11928658
- [Background] Risser NL, Belcher DW. Adding spirometry, carbon monoxide, and pulmonary symptom results to smoking cessation counseling: a randomized trial. J Gen Intern Med. 1990 Jan-Feb;5(1):16-22. doi: 10.1007/BF02602303. PMID 2405112
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh/68016540
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh/68011320
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh?term=spirometry